CLINICAL TRIAL: NCT06795984
Title: Is There a Correlation Between Endometrial CD56 Levels and the Unfavorable KIR AA Genotype in IVF Implantation Success?
Status: Completed | Type: Observational
Sponsor: Calla IVF Center (Other)
Responsible Party: Sponsor
Other Study IDs: CALLAIVF KIR HLAC
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Rate IVF; Blastocyst IVF

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KIR AA (Group A): In any pregnancy, the maternal KIR genotype could be AA (mostly inhibitory KIRs), AB, or BB (mostly activating KIRs). A KIR AA haplotype is defined as cen-A and tel-A
  Interventions: Other: Establishing the correlation between KIR AA and KIR non-AA and CD56 endometrial cells and IVF succes
- KIR non AA (Group B): In any pregnancy, the maternal KIR genotype could be AA (mostly inhibitory KIRs), AB, or BB (mostly activating KIRs). KIR Bb haplotype is described as cenB/telB, cenA/telB, or cenB/telA
  Interventions: Other: Establishing the correlation between KIR AA and KIR non-AA and CD56 endometrial cells and IVF succes

INTERVENTIONS:
Other: Establishing the correlation between KIR AA and KIR non-AA and CD56 endometrial cells and IVF succes — The analysis aimed to compare CD56 levels between patients with the KIR AA genotype and those without. A multiple linear regression model was used to determine the predictive value of CD56+ levels, KIR genotype, and age on the number of blastocysts.

SUMMARY:
This prospective observational study was conducted over 12 months and involved 80 IVF patients aged 20-40 years. Patients were divided into two groups based on KIR genotype (KIR AA and non-KIR AA). Endometrial biopsies were collected during the mid-luteal phase for immunohistochemical analysis of CD56+ NK cell levels. Statistical analyses, including logistic regression and ROC curve evaluation, assessed the relationship between CD56 levels, KIR genotype, and implantation success.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 20-40 years.
* Normal uterine cavity confirmed by hysteroscopy or sonohysterography.
* At least three previous failed IVF cycles or a history of recurrent pregnancy loss (RPL).

Exclusion Criteria:

* uterine abnormalities,
* systemic autoimmune diseases,
* severe male infertility factors.

Ages: 21 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — females undergoing IVF with endometrial biopsy for CD56
Study Population: A total of 80 patients were included, with 40 in each group (KIR AA and non-KIR AA). All participants provided written informed consent, and the study protocol was approved by the institutional ethics committee.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
the relationship between endometrial CD56+ NK cells, KIR AA genotypes, and IVF success. | 12 months
  The value of CD56 NK cell and KIR AA in patients undergoing IVF and pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Calla Ivf Center, Oradea, Bihor County, Romania